CLINICAL TRIAL: NCT06363279
Title: Validation of the French Translation of the Affinity for Technology Interaction (ATI) Scale Questionnaire and Assessment of the Predisposition of Healthy Adults and Stroke Survivors to Use Technological Tools in Rehabilitation.
Brief Title: Validation of the French ATI Scale and Predisposition to Use Technological Tools in Rehabilitation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024/24JAN/044
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaires on predisposition to the use of technology (Other): The questionnaire is divided into 4 main sections:
  * General information: Questions on age, gender, postal code, country, socio-professional status and level of education.
  * ATI questionnaire in French: Questionnaire consisting of 9 items to assess affinity for interaction with technological systems (such as mobile phones, computers, television, etc.).
  * Face validity and perceived usefulness: Five statements designed to assess the face validity and perceived usefulness of the questionnaire to respondents. The response options for each statement are in the form of a Likert scale ranging from 'strongly disagree' to 'strongly agree'.
  * Predisposition to use technology: Questionnaire to assess predisposition to use new technologies in general and specifically in telerehabilitation.
  Interventions: Other: Conducting questionnaires

INTERVENTIONS:
Other: Conducting questionnaires — The questionnaires will be administered online or in person.

SUMMARY:
Aim of the study: The first aim of this study is to validate the translation of the Affinity for Technology Interaction (ATI) questionnaire. This questionnaire was developed in English by Franke, Attig and Wessel in 2019. It consists of 9 items and was developed to assess a person's tendency to actively engage in technological interaction, or the ease with which a person uses technological tools. Currently, the questionnaire has been translated into French by our research team according to good practice recommendations, but this French version has not yet been validated. To validate the translation of a questionnaire, it is necessary to have it completed by a large number of subjects from the population of interest. In neurorehabilitation, measuring this affinity will make it possible to better identify patients who are more likely to adhere to tele-rehabilitation and thus direct them towards this type of treatment as a complement to conventional rehabilitation.

The second objective is to determine the extent to which the general population is prepared to use technological tools as part of their rehabilitation. The aim is to gain a better understanding of the profile of people who could potentially benefit from tele-rehabilitation. Accessibility to the technologies, their expectations and barriers will also be explored as part of this study.

DETAILED DESCRIPTION:
The primary objective of this cross-sectional study is to validate the French translation of the "Affinity for Technology Interaction" questionnaire in the general adult population and in an adult population that has suffered a stroke.

The secondary objective is to assess the propensity of these populations to use technological tools in everyday life and in rehabilitation.

The experiment is a cross-sectional study (online and paper survey). Subjects will be recruited in two ways: 1) via the Cliniques universitaires Saint-Luc; 2) via posters/flyers in paper and digital formats, the Internet (social networks), public places (university, etc.), acquaintances of the participants and of the research team, and via colleagues of the doctors/physiotherapists (samples of convenience and "snowballing"). Posters and publications on social networks will include information about the experiment and a link to the online questionnaire.

People who want to take part in the online survey will have to click on the link to be directed to the questionnaire on REDCap. Once they have given their consent electronically, i.e. by ticking 'yes' to 'I agree to take part in this study of my own free will', the questionnaire will appear and participants will be able to complete it (this will take approximately 5-10 minutes). Once they have completed the questionnaire, their participation in the study will be terminated. The questionnaire will be available online for a period of 12 months.

For people who wish to take part in the paper survey, after signing the information and consent documents, they will complete the paper version of the questionnaire with the assistance of an investigator. Once the questionnaire has been completed, their participation in the study will be terminated.

Selection criteria for subjects to be included in the experiment (all randomly selected subjects, all evaluable subjects, etc.).

- Healthy subjects: The healthy subjects included in the study will be volunteers recruited either through the Saint-Luc University Hospitals or through social networks, but also in public places (university), as well as through fellow physiotherapists and doctors. This study will be offered in several French-speaking countries (France, Canada, Belgium).

- People who have had a stroke: Stroke survivors enrolled in the study will be volunteers recruited either through the Saint-Luc University Hospitals Physical Medicine and Rehabilitation Department or through social networks and public places.

Precise statement of the main data to be evaluated during the experiment. The questionnaire (see appendix) is divided into 4 main sections: general information; French version of the ATI questionnaire; face validity and perceived usefulness; predisposition to use new technologies.

* General information: Questions on age, gender, postal code, country, socio-professional status and level of education. These data will be used to describe the sample studied (descriptive statistics) and to obtain the information needed to determine the factors associated with the ATI questionnaire score in multiple linear regression analyses. For post-stroke subjects, the questionnaire will be completed with information on the date of stroke, its functional classification, Rankin score and MOCA.
* French version of the ATI questionnaire: Questionnaire consisting of 9 items designed to assess the affinity for interaction with technological systems (such as mobile phones, computers, television, etc.). The response options for each item are in the form of a Likert scale ranging from "strongly disagree" (= 1) to "strongly agree" (= 6). A total score including the 9 items is then calculated to obtain the subject's score.
* Face validity and perceived usefulness: Five statements designed to assess the face validity and perceived usefulness of the questionnaire to respondents. The response options for each statement are in the form of a Likert scale ranging from 'strongly disagree' to 'strongly agree'.
* Predisposition to use technology: Questionnaire to assess predisposition to use new technologies in general and specifically in telerehabilitation. This questionnaire includes questions about the rehabilitation that the subjects are currently undergoing (type, frequency, investment and difficulties of access), as well as their propensity to use new tools (in rehabilitation and in daily life).

Expected duration of subjects' participation. The duration of participation includes only the time needed to complete the questionnaire. Without a break, we estimate that it will take about 10 minutes to complete the questionnaire. After that, participation in the study is over.

Data analysis methods including missing, unused or erroneous data. REDCap software will be used to conduct the surveys. REDCap is a statistical survey and online form creation software. It allows questionnaires to be published on the web or on smartphones to collect data. The software allows anonymous participation and an unlimited number of participants and questions. We can choose the start and end dates for the survey, as well as a server location for secure data storage. Thanks to this software, data collection will take place in real time and we will be able to monitor the results.

We will also be able to obtain the results of the survey in the form of statistics or graphs (e.g. number of responses per question) at any time. The survey results will be exported anonymously and securely in various formats (Excel, CSV, PDF, etc.) for processing and analysis in statistical software.

The data collected via the paper version (mainly for stroke patients) and REDCap will be imported into Excel and analysed using SPSS and R. The face validity, perceived usefulness and other aspects such as the ergonomics of the questionnaire will be assessed via the statements at the end of the questionnaire and the time taken to complete the questionnaire. We will also assess the reliability of the questionnaire by calculating its internal consistency (Cronbach Alpha) and its dimensionality by calculating the number of dimensions (exploratory factorial analysis).

Multiple linear regression analyses will also be carried out to assess the association between certain variables (e.g. age) and the score on the ATI questionnaire. Results are presented as coefficients with their 95% confidence intervals. All p-values are two-tailed and the significance level is set at p = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (> 18 years)
* Speak and understand French;
* Be able to give consent in paper or electronic format.
* Have had a single stroke;
* Have been out of hospital for at least 1 month.

Exclusion Criteria:

* Severe comprehension problems ;
* Inability to complete the questionnaire;
* Severe comprehension problems, prior to or following the stroke, preventing planned assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
ATI - affinity technology interaction scale | Baseline
  Evaluation scale in the form of a self-questionnaire to assess a person's affinity with technological communication tools.
  French version of the ATI questionnaire: Questionnaire consisting of 9 items designed to assess the affinity for interaction with technological systems (such as mobile phones, computers, television, etc.). The response options for each item are in the form of a Likert scale ranging from "strongly disagree" (= 1) to "strongly agree" (= 6). A total score including the 9 items is then calculated to obtain the subject's score.

SECONDARY OUTCOMES:
Scale for assessing a person's readiness to use technological tools as part of their rehabilitation | Basline
  Self-questionnaire concerning people's habits in relation to the use of technological tools, both overall and more specifically in terms of healthcare.
  Predisposition to use technology: Questionnaire to assess predisposition to use new technologies in general and specifically in telerehabilitation. This questionnaire includes questions about the rehabilitation that the subjects are currently undergoing (type, frequency, investment and difficulties of access), as well as their propensity to use new tools (in rehabilitation and in daily life).

CONTACTS AND LOCATIONS:
Overall Officials: Lejeune Thierry, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Clinique Universitaires Saint-Luc, Brussels, Woluwé-Saint-Lambert, Belgium